CLINICAL TRIAL: NCT01631435
Title: Evaluation of the PillCam® Platform With the PillCam Crohn's Disease Capsule in Visualization of Lesions in the Small Bowel and Colon That May Indicate Crohn's Disease
Brief Title: PillCam® Platform With the PillCam Crohn's Disease Capsule
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MA-206
Record Dates: First submitted 2012-06-28; First posted 2012-06-29 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2015-03

CONDITIONS: Crohn's Disease
Keywords: All subjects will have evidence of active symptoms associated with Crohn's disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bowel prep regimen (Other): Each study subject will undergo a bowel preparation followed by a PillCam procedure.
  Interventions: Other: Pillcam colon capsule and PillCam™ Prep Procedure; Device: Ileocolonoscopy

INTERVENTIONS:
Other: Pillcam colon capsule and PillCam™ Prep Procedure — PillCam® Crhon capsule preparation will include a clear liquid diet and administration of a purgative sulfate-free polyethylene glycol electrolyte lavage (SF-ELS) solution (e.g. Nulytely) divided into two doses: the first dose on the evening before the exam and the 2nd dose on the morning of the exam day.
Device: Ileocolonoscopy — Conventional ileocolonoscopy Examination (same day or within 24 hours)of CE procedure
  • Ileocolonoscopy with intubation of terminal ileum

SUMMARY:
This is a prospective, multi-center (up to 6 sites) study which aims to To establish the effectiveness of the PillCam Platform with the PillCam Crohn's capsule as demonstrated by visualizing the small bowel and colon in patients with active symptoms associated with Crohn's disease (CD).

DETAILED DESCRIPTION:
This is a prospective, multi-center (up to 6 sites) study which aims to evaluate the diagnostic yield and safety of the PillCam Platform with the CD capsule in subjects with symptoms associated with Crohn's disease. All subjects to be enrolled in this study will have evidence of active symptoms associated with Crohn's disease. Each subject will be required to follow a bowel preparation regimen and will undergo the Crohn's Disease capsule endoscopy procedure and thereafter the ileocolonoscopy procedure on the same day. The ileocolonoscopy procedure may be done the following day per physician discretion. If the ileocolonoscopy procedure is done within 24 hours from the CE procedure, the subject will stay on clear liquid diet. Observations/ assessments to be conducted in the trial detailed in the sections below:

Visit 1; Screening visit

* Informed consent process
* screening for eligibility to participate in the study
* Inclusion/exclusion criteria
* Small bowel patency test
* Demographic data
* Pregnancy test
* General medical history

Visit 2; PillCam® Crohn's capsule ingestion

* PillCam® CD bowel preparation
* Capsule endoscopy Conventional ileocolonoscopy Examination (same day or within 24 hours)
* Ileocolonoscopy with intubation of terminal ileum

Follow up period (5-9 days following visit 2)

• CE Follow up telephone contac

ELIGIBILITY:
Inclusion Criteria:

1. Subject ages 18-75 years, inclusive
2. Subject has known CD and signs and symptoms of active disease including one of the following:

   * Chronic diarrhea
   * Chronic abdominal pain
   * Rectal bleeding
3. Subject has at least one of the following within three months of enrollment:

   * Positive inflammatory marker (ESR, CRP, thrombocytosis, leukocytosis, fecal lactoferrin, fecal alpha-1 antitrypsin)
   * Anemia (hemoglobin level below normal reference range)
   * Hypoalbuminemia (albumin below normal reference range)
   * Weight loss
4. Proven patency by the Agile capsule or another approach deemed clinically acceptable by the investigator, e.g. CT enterography, performed within the 90 days prior to enrollment.
5. Subject agrees to sign consent form

Exclusion Criteria:

1. Indeterminate Colitis
2. Ulcerative Colitis
3. Antibiotic Associated Colitis
4. Stool positive for Ova &Parasite and for Clostridium difficile toxin within 3 months of enrollment
5. Other known infectious cause of increased symptoms
6. Known history of intestinal obstruction or current obstructive symptoms, such as severe abdominal pain with accompanying nausea or vomiting, based on investigator judgment.
7. Definite long stricture seen on radiological exam.
8. Non-steroidal anti-inflammatory drugs including Aspirin, (twice weekly or more) during the 4 weeks preceding enrollment
9. Suspected GI stricture, followed by Pillcam Patency study or other imaging study that could not prove patency of the GI tract.
10. Subject has had prior abdominal surgery of the gastrointestinal tract in the last 6 months, other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator.
11. Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
12. Subjects with known or suspected delayed gastric emptying
13. Subjects with known or suspected delayed Small bowel motility
14. Subject suffers from any condition, such as swallowing problems, which precludes compliance with study and/or device instructions.
15. Subject has Type I or Type II Diabetes.
16. Subject has any allergy or other known contraindication to the medications used in the study.
17. Subject has any condition, which precludes compliance with study and/or device instructions.
18. Women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
19. Concurrent participation in another clinical trial using any investigational drug or device.
20. Subject suffers from a life threatening condition.
21. Subject with a history or clinical evidence of renal disease and/or previous clinically significant laboratory abnormalities of renal function parameters.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-06; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debbra Helper, MD, Principal Investigator — Indiana University, Indianapolis , USA
Locations (1):
- IU School of Medicine - Gastroenterology, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: total of 39 cases have been excluded and were not enrolled to the study due to the follwoings: 38 cases are screen faliure
  1 case due to physican decision - the patient not eligible for the study
Groups:
- Bowel Prep Regimen: Each study subject will undergo a bowel preparation followed by a PillCam procedure.
  Pillcam colon capsule and PillCam™ Prep Procedure: PillCam® Crhon capsule preparation will include a clear liquid diet and administration of a purgative sulfate-free polyethylene glycol electrolyte lavage (SF-ELS) solution (e.g. Nulytely) divided into two doses: the first dose on the evening before the exam and the 2nd dose on the morning of the exam day.
  Ileocolonoscopy: Conventional ileocolonoscopy Examination (same day or within 24 hours)of CE procedure
  • Ileocolonoscopy with intubation of terminal ileum
Period: Overall Study
Arm/Group | Bowel Prep Regimen
Started | 75
Completed | 66
Not Completed | 9
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — incomplete study procedure | 5

BASELINE CHARACTERISTICS:
Arm/Group | Bowel Prep Regimen
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 65
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.94 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 53
  Israel | 13

OUTCOME MEASURES:

1. Primary Outcome: Per-subject Diagnostic Yield of the PillCam Platform With the CD Capsule Within the Terminal Ileum and Colon as Compared to the Ileocolonoscopy Diagnostic Yield Within the Terminal Ileum and Colon
Description: the primary outcome will be evalluated as follow: The number of subjects having active Crohn's disease in their terminal ileum and / or colon as detected by the PillCam Platform with the CD capsule and ileocolonoscopy.
  The analysis related to the primary endpoint was applied for the terminal ileum and colon only due to the limited access of ileocolonoscopy.
  Each patient was classified as follows:
  * Active Crohn's disease is likely
  * Active Crohn's disease is NOT likely "Active Crohn's disease" included the followings lesions:
  * Aphthous ulceration
  * Ulcers (other than Aphthous)
  * Bleeding
  * Inflammatory stricture Lesions other than the above list were classified as "Non active Crohn's disease."
Time Frame: All the end points and outcomes measures will be evaluated within 4 months from end of enrollment
Population: subjects with symptoms associated with Crohn's disease
Measure: Number; unit: number of subjects
Groups:
- # Casesclassified as "Active CD is Likely" by CE: The number of subjects having active Crohn's disease(CD) in their TI and / or colon as detected by the PillCam Platform with the CD capsule endoscopy(CE).
  "Active Crohn's disease" included the followings lesions:
  * Aphthous ulceration
  * Ulcers (other than Aphthous)
  * Bleeding
  * Inflammatory stricture Lesions other than the above list were classified as "Non active Crohn's disease."
- # Casesclassified as "Active CD is Likely" by IC: The number of subjects having active Crohn's disease(CD) in their TI and / or colon as detected by the PillCam Platform with the Ileo colonoscopy (IC) procedure.
  "Active Crohn's disease" included the followings lesions:
  * Aphthous ulceration
  * Ulcers (other than Aphthous)
  * Bleeding
  * Inflammatory stricture Lesions other than the above list were classified as "Non active Crohn's disease."
Arm/Group | # Casesclassified as "Active CD is Likely" by CE | # Casesclassified as "Active CD is Likely" by IC
Number analyzed (Participants) | 66 | 66
number of subjects | 55 | 46

ADVERSE EVENTS:
Arm/Group | Bowel Prep Regimen
Serious Adverse Events (participants affected / at risk) | 3/66
Other Adverse Events (participants affected / at risk) | 11/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bowel Prep Regimen (N=66)
Bowel preparation (Gastrointestinal disorders) | 1 (1) — One case of hospitalization due to abdominal pain related to preparation (CE and IC procedure were not done)
CE Proceudre (Gastrointestinal disorders) | 1 (1) — o One case of hospitalization and medical intervention due to abdominal pain related to the CE procedure due to bowel obstruction
patency capsule (Gastrointestinal disorders) | 1 (1) — One case of hospitalization and medical intervention due to Abdominal pain, nausea, vomiting, blotting and fever related to the ingestion of the
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Bowel Prep Regimen (N=66)
nausea duo to colon preparation (Gastrointestinal disorders) | 11/11 (11) — nausea
vomiting due to colon preparation (Gastrointestinal disorders) | 6 (6)
mild headache due to colon preparation (Gastrointestinal disorders) | 1 (1)
mild abdominal cramping (Gastrointestinal disorders) | 1 (1) — due to colon preparation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No